CLINICAL TRIAL: NCT04800471
Title: Improving Glycemic Control and Clinical Outcomes in DM2 Patients in the Ambulatory Setting, a Pilot Study
Brief Title: Improving Glycemic Control in DM2 Patients in the Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ilias Spanakis, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00095543
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Smart insulin pens and CGM (Active Comparator): Participants in this group will be monitored by Smart Insulin pens and Continuous Glucose Monitoring Devices
  Interventions: Device: Smart insulin pens and CGM
- Point of Care Glucose Group (Placebo Comparator): Participants in this group will be monitored by point of care glucose values
  Interventions: Other: Point of Care Glucose Group

INTERVENTIONS:
Device: Smart insulin pens and CGM — Participants in this group will be monitored by Smart Insulin pens and Continuous Glucose Monitoring Devices
  Arms: Smart insulin pens and CGM
Other: Point of Care Glucose Group — Participants in this group will be monitored by POC glucose values.
  Arms: Point of Care Glucose Group

SUMMARY:
More than 10.5% of the US population has diabetes mellitus. The objective of this pilot study is to evaluate whether smart insulin pens combined with CGM devices can improve glucose control in patients with type 2 diabetes (T2D)

DETAILED DESCRIPTION:
Diabetes is affecting millions of Americans. High glucose levels lead to complications such as heart attacks, stroke or blindness. Patients with diabetes need to exercise at least 150 min/week, a goal however that is not usually achieved. Reducing high glucose levels may unfortunately lead to very low glucose values-hypoglycemia, a condition that can lead to loss of consciousness or even death. Both of these conditions, high and low glucose levels, can therefore lead to visits to the Emergency department or hospitalizations. In fact, patients with diabetes have frequent admissions to the hospital. Additionally, many of them are admitted again, immediately or in less than 30 days after hospital discharge. Most of patients with diabetes are monitoring their glucose values with finger-stick glucose testing. Continuous Glucose Monitors (CGMs) are new devices that can monitor glucose continuously (every couple of minutes) without the need of finger-stick glucose testing. Similar to the glucometers, CGM devices can record glucose values, which can then be obtained by the clinicians, who can help them to modify DM medications. In addition to using CGM devices for diabetes management, smart insulin pens can be used in order to help with diabetes control. These devices can store and transfer data to the medical doctors, making them aware about the patients' glucose values. Moreover there are different health solutions available to manage patients including mobile health and telemedicine, which can help combining and transferring these data remotely. Briefly, telemedicine is a way to deliver healthcare where providers and patients communicate through alternative methods (telephone or other electronic method for example) instead of only traditional in-person office visits. Using telemedicine to replace some routine office visits can improve access to healthcare. It can also improve communication between patients and providers which is often a challenge to diabetes management. You may be able to more quickly and safely change medications to help the patients' diabetes control.

In this application we are going to examine whether utilizing telemedicine is a better communication tool between patients and providers and if it will lead to improved blood sugar control and increased exercise pattern compared to traditional monitoring with glucometers and in-person office visits only. We believe that this intervention may lead to better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Insulin-treated patients with DM2 (treated with basal-bolus insulin regimens (MDI), ± non-insulin medications) and Uncontrolled glycemic control

Exclusion Criteria:

* History of type 1 DM (DM1)
* Pregnant Patients
* Extensive skin changes/disease or allergies that preclude wearing the CGM sensor
* Subjects who have end-stage renal disease requiring dialysis
* Significant psychiatric illness or any other condition rendering the subject incapable of understanding the objectives and potential consequences of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Started | 15 | 15
Completed | 11 | 13
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — The average age for each group
  years | 65.00 (7.05) | 63.91 (8.68) | 64.50 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Total males and females in each group
  Participants
    Female | 0 | 2 | 2
    Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race counts in each group
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 8 | 16
    White | 3 | 5 | 8
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] — Average Baseline HbA1c per group
  percentage of HbA1c | 9.47 (1.57) | 9.37 (1.18) | 9.42 (1.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hyperglycemia (Percent Change in HbA1c)
Description: HbA1C test is a blood test that shows your average level of blood glucose, also called blood sugar, over the past three months.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: HbA1c percent change
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
HbA1c percent change | -2.2 ((-3.1, -1.3)) [-3.1 to -1.3] | -1.0 ((1.9, -0.13) [-1.9 to -0.13]

2. Secondary Outcome: Change in Hyperglycemia (Percent Change in HbA1c)
Description: The change in Hb1Ac (baseline to 6 months) is reported in percent
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: HbA1c percent change
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
HbA1c percent change | -2.2 [-3.2 to -1.3] | -1.1 [-2.0 to -0.2]

3. Secondary Outcome: Change in Hypoglycemia
Description: Change in hypoglycemic episodes (CGM glucose <70 mg/dl for at least 15 min)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Hypoglycemic events <70 mg/dL
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Hypoglycemic events <70 mg/dL | 0.6 [-2.2 to 1] | -1.5 [-3.0 to -0.1]

4. Secondary Outcome: Change in Hypoglycemia
Description: Change in hypoglycemic episodes (CGM glucose <70 mg/dl for at least 15 min)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Hypoglycemia events < 70 mg/dL
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Hypoglycemia events < 70 mg/dL | 0.5 [-1.1 to 2.1] | -0.1 [-1.6 to 1.4]

5. Secondary Outcome: Change in Clinically Significant Hypoglycemia
Description: Change in clinically significant hypoglycemic episodes (CGM<54 mg/dl at least 15 min)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Hypoglycemic events <54mg/dL
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Hypoglycemic events <54mg/dL | 0.1 [-0.8 to 0.9] | 0.0 [-0.8 to 0.8]

6. Secondary Outcome: Change in Clinically Significant Hypoglycemia
Description: Change in clinically significant hypoglycemic episodes (CGM<54 mg/dl at least 15 min)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Hypoglycemic events <54mg/dL
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Hypoglycemic events <54mg/dL | 0.1 [-0.8 to 0.9] | -0.5 [-1.3 to 0.2]

7. Secondary Outcome: Change in Percentage of Glucose Values in Range (70-180 mg/dl)
Description: We report the change of percentage of CGM glucose values in the range (70-180 mg/dl)
Time Frame: up to 3 months
Measure: Mean (95% Confidence Interval); unit: Change in Percentage of glucose values
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Change in Percentage of glucose values | 13.4 [-8.6 to 35.5] | 13.7 [-6.6 to 34.0]

8. Secondary Outcome: Change in Percentage of Glucose Values in Range (70-180 mg/dl)
Description: We report the change of percentage of CGM glucose values in the range (70-180 mg/dl)
Time Frame: up to 6 months
Measure: Mean (95% Confidence Interval); unit: Change in Percentage of glucose values
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Change in Percentage of glucose values | 15.4 [-6.7 to 37.4] | 17.3 [-3.0 to 17.5]

9. Secondary Outcome: Change in Percentage of Glucose Values Below Range (<70 mg/dl)
Description: We report the change of percentage of CGM glucose values below the range (<70 mg/dl)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Change in Percentage of glucose values
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Change in Percentage of glucose values | 0.1 [-0.8 to 1.0] | -0.2 [-1.1 to 0.6]

10. Secondary Outcome: Change in Percentage of Glucose Values Below Range (<70 mg/dl)
Description: We report the change of percentage of CGM glucose values below the range (<70 mg/dl)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Change in Percentage of glucose values
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Change in Percentage of glucose values | 0.4 [-0.5 to 1.3] | -0.9 [-1.7 to -0.1]

11. Secondary Outcome: Change in Percentage of Glucose Values Above Range (>180 mg/dl)
Description: We report the change of percentage of CGM glucose values Above Range (>180 mg/dl)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Change in Percentage of glucose values
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Change in Percentage of glucose values | -10.4 [-11.1 to -0.8] | -16.2 [-35.1 to -2.6]

12. Secondary Outcome: Change in Percentage of Glucose Values Above Range (>180 mg/dl)
Description: We report the change of percentage of CGM glucose values Above Range (>180 mg/dl)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Change in Percentage of glucose values
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
Change in Percentage of glucose values | -20.4 [-40.9 to 0.03] | -17.9 [-36.7 to 0.9]

13. Secondary Outcome: Change in Glucose Variability
Description: Change in Coefficient of Variation (CV)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: percentage of coefficient of variation
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
percentage of coefficient of variation | 1.9 [-4.4 to 8.1] | -1.7 [-7.4 to 4.1]

14. Secondary Outcome: Change in Glucose Variability
Description: Change in Coefficient of Variation (CV)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of coefficient of variation
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
Number analyzed (Participants) | 11 | 13
percentage of coefficient of variation | -2.0 [-8.3 to 4.2] | -3.0 [-8.7 to 2.8]

ADVERSE EVENTS:
Time Frame: From enrollment to 6 months
Arm/Group | Smart Insulin Pens and CGM | Point of Care Glucose Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT04800471/Prot_SAP_005.pdf
  • Informed Consent Form (2023-02-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT04800471/ICF_006.pdf